CLINICAL TRIAL: NCT05293145
Title: AVANCE-Houston Building Futures Healthy Marriage and Responsible Fatherhood Program Evaluation
Brief Title: AVANCE-Houston Building Futures Program Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/33
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Youth

STUDY DESIGN:
Intervention Model Description: Primary Services Participants receive 14 hours of Survival Skills for Healthy Families curricula delivered over a series of 7 weekly workshops, or 16 hours of Survival Skills for Healthy Families curricula delivered over one weekend followed by 2 hours of a Reflections Workshop delivered two weeks later. Participants also receive support services delivered by Family Coaches and Career Coaches as needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Building Futures Program Primary Services (Experimental): Primary Services Participants receive 14 hours of Survival Skills for Healthy Families curricula delivered over a series of 7 weekly workshops. Participants also receive support services delivered by Family Coaches and Career Coaches as needed.
  Interventions: Other: Building Futures Program Primary Services

INTERVENTIONS:
Other: Building Futures Program Primary Services — Primary Services Participants receive 14 hours of Survival Skills for Healthy Families curricula delivered over a series of 7 weekly workshops. Participants also receive support services delivered by Family Coaches and Career Coaches as needed.

SUMMARY:
AVANCE seeks to understand if participation in the AVANCE-Houston Building Futures (A-HBF) program is associated with improved outcomes among the target population of at-risk, homeless, and incarcerated youth. Additionally, the evaluation will examine how and why participant-level characteristics such as relationship status, life status, and demographics are associated with greater or lesser benefit from A-HBF program participation. This research will provide insights about the Survival Skills for Healthy Families curriculum and its effectiveness for the target population that can be used in the development of future programming efforts.

DETAILED DESCRIPTION:
Trauma-informed services are needed to improve self-sufficiency, economic stability, and healthy relationships among at-risk, homeless, and incarcerated youth in Harris County, especially those living in areas with high numbers of single-family households, high poverty rates, low educational attainment, high teen pregnancy rates, high incidence of domestic violence, and high involvement with the (juvenile) justice system. AVANCE-Houston's Building Futures program (A-HBF) aims to facilitate successful transitions to adulthood for cohorts of at-risk and homeless youth by offering healthy relationship and marriage education through the Survival Skills for Healthy Families (SSHF) curriculum.

Developed by Family Wellness Associates, SSHF is an evidence-based curriculum delivered through a series of workshops that focus on communication skills, conflict resolution, knowledge of the benefits of marriage, stress and anger management, parenting skills, financial literacy, job and career advancement, and relationship skills to improve family and economic stability. AVANCE will offer the curriculum via weekly workshops for youth that take place in targeted high-need areas.

AVANCE seeks to understand if participation in the A-HBF program is associated with improved outcomes among the target population of at-risk and homeless youth. Additionally, the evaluation will examine how and why participant-level characteristics such as relationship status, life status, and demographics are associated with greater or lesser benefit from A-HBF program participation. This research will provide insights about the SSHF curriculum and its effectiveness for the target population that can be used in the development of future programming efforts.

ELIGIBILITY:
Inclusion Criteria:

* Youth (aged 14-18)
* High-needs school districts enrolled in grades 9-12
* Residing in juvenile detention center

Exclusion Criteria:

* Adult (age 18 and older)
* Youth (age 14 and younger)
* Not enrolled in school (non-incarcerated youth)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 718 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Healthy partner relationship behavior measurement #1 | Change from baseline in partner relationship behavior from enrollment to 12-month follow-up
  1A) Will participants report healthier partner relationship behaviors after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  5 items - levels of reported skill with key relationship behaviors (categories; 4-point scale)
  Measured on the Healthy Parenting Behavior Scale #1 as:
  1=I am extremely good at this, 2=I am good at this, 3=I am bad at this, 4=I am extremely bad at this
  The lower the rating, the better the score.
Healthy partner relationship behavior measurement #2 | Change from baseline in partner relationship behavior from enrollment to 12-month follow-up
  1B) Will participants report healthier partner relationship behaviors after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  6 items - frequency of engagement in key relationship behaviors (categories; 5-point scale)
  Measured on the Healthy Parenting Behavior Scale #2 as:
  1=none of the time, 2=some of the time, 3=half of the time, 4=most of the time, 5=all of the time The higher the rating, the better the score for 1 item. 5 items are reverse scored, with the lower the rating, the better the score.

SECONDARY OUTCOMES:
Healthy partner relationship attitudes measurement #1 | Change from baseline in partner relationship attitudes to immediately after program completion
  2A) Will participants report healthier partner relationship attitudes after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  9 items - levels of agreement with relationship beliefs (categories; 4-point scale)
  Measured on the Healthy Relationship Attitudes Scale #1 as:
  1=strongly agree, 2=agree, 3=disagree 4=strongly disagree The higher the rating, the better the score for 7 items. 2 items are reverse scored, with the lower the rating, the better the score.
Healthy partner relationship attitudes measurement #2 | Change from baseline in partner relationship attitudes to immediately after program completion
  2B) Will participants report healthier partner relationship attitudes after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  3 items - likelihood of key relationship beliefs (categories; 5-point scale)
  Measured on the Healthy Relationship Attitudes Scale #2 as:
  1=almost no chance, 2=some chance but probably not, 3=a 50-50 chance, 4=a good chance, 5=almost certain The higher the rating, the better the score for 1 item. 2 items are reverse scored, with the lower the rating, the better the score.
Healthy sexual attitudes measurement #1 | Change from baseline in sexual attitudes from enrollment to immediately after program completion
  3A) Will participants report healthier sexual attitudes after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  7 items - levels of agreement with key sexual attitudes (categories; 4-point scale)
  Measured on the Healthy Sexual Attitudes Scale #1 as:
  1=strongly agree, 2=agree, 3=disagree 4=strongly disagree The higher the rating, the better the score for 3 items. 4 items are reverse scored, with the lower the rating, the better the score.
Healthy financial attitudes measurement #1 | Change from baseline in financial attitudes from enrollment to 12-month follow-up
  4A) Will participants report healthier financial attitudes after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  8 items - levels of agreement with key financial attitudes (categories; 5-point scale)
  Measured on the Healthy Financial Attitudes Scale #1 as:
  1=strongly disagree, 2=disagree, 3=neither agree or disagree, 4=agree, 5=strongly agree
Healthy employment attitudes measurement #1 | Change from baseline in employment attitudes to immediately after program completion
  5A) Will participants report healthier employment attitudes after they complete primary services and support services in the AVANCE-Houston Building Futures Program?
  Items measured include:
  8 items - levels of agreement with key employment attitudes (categories; 5-point scale)
  Measured on the Healthy Employment Attitudes Scale #1 as:
  1=strongly disagree, 2=disagree, 3=neither agree or disagree, 4=agree, 5=strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- AVANCE-Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.